CLINICAL TRIAL: NCT06724406
Title: FAMily-centered WEight Loss for Black Adults (FAM WEL B-ing): Optimization and Evaluation Using Multiphase Optimization Strategy (MOST) and Social Network Analysis (SNA)
Brief Title: FAMily-centered WEight Loss for Black Adults (FAM WEL B-ing)
Acronym: FAM WEL B-ing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 24-1302; R61HL169357 (NIH)
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Obesity and Overweight; Diabetes Mellitus; Weight Loss; Behavior Change
Keywords: weight loss program; African American or Black families; nutrition and physical activity behavior change
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Session 5, In-Person, Communication and Cohesion (Experimental): Participants will receive core behavioral weight loss group sessions and 5 family skills training sessions in-person with content covering communication and cohesion
  Interventions: Behavioral: Family Skills Training Session Quantity: 5; Behavioral: Family Skills Training Session Mode: In-person; Behavioral: Family Skills Training Content: Communication; Behavioral: Family Skills Training Content: Cohesion
- Session 5, In-Person, Communication and No Cohesion (Experimental): Participants will receive core behavioral weight loss group sessions and 5 family skills training sessions in-person with content covering communication but no cohesion
  Interventions: Behavioral: Family Skills Training Session Quantity: 5; Behavioral: Family Skills Training Session Mode: In-person; Behavioral: Family Skills Training Content: Communication; Behavioral: Family Skills Training Content: No Cohesion
- Session 5, In-Person, Cohesion and No Communication (Experimental): Participants will receive core behavioral weight loss group sessions and 5 family skills training sessions in-person with content covering cohesion but no communication
  Interventions: Behavioral: Family Skills Training Session Quantity: 5; Behavioral: Family Skills Training Session Mode: In-person; Behavioral: Family Skills Training Content: Cohesion
- Session 5, In-Person, No Communication and No Cohesion (Experimental): Participants will receive core behavioral weight loss group sessions and 5 family skills training sessions in-person with content covering no communication but no cohesion
  Interventions: Behavioral: Family Skills Training Session Quantity: 5; Behavioral: Family Skills Training Session Mode: In-person; Behavioral: Family Skills Training Content: Communication; Behavioral: Family Skills Training Content: Cohesion; Behavioral: Family Skills Training Content: No Communication
- Session 5, On-Line, Communication and Cohesion (Experimental): Participants will receive core behavioral weight loss group sessions and 5 family skills training sessions on-line with content covering communication and cohesion
  Interventions: Behavioral: Family Skills Training Session Quantity: 5; Behavioral: Family Skills Training Content: Communication; Behavioral: Family Skills Training Content: Cohesion; Behavioral: Family Skills Training Session Mode: Online
- Session 5, On-Line, Communication and No Cohesion (Experimental): Participants will receive core behavioral weight loss group sessions and 5 family skills training sessions on-line with content covering communication but no cohesion
  Interventions: Behavioral: Family Skills Training Session Quantity: 5; Behavioral: Family Skills Training Content: Communication; Behavioral: Family Skills Training Session Mode: Online; Behavioral: Family Skills Training Content: No Cohesion
- Session 5, On-Line, Cohesion and No Communication (Experimental): Participants will receive core behavioral weight loss group sessions and 5 family skills training sessions on-line with content covering cohesion but no communication
  Interventions: Behavioral: Family Skills Training Session Quantity: 5; Behavioral: Family Skills Training Content: Cohesion; Behavioral: Family Skills Training Session Mode: Online; Behavioral: Family Skills Training Content: No Communication
- Session 5, On-Line, No Communication and No Cohesion (Experimental): Participants will receive core behavioral weight loss group sessions and 5 family skills training sessions on-line with content covering no communication and no cohesion
  Interventions: Behavioral: Family Skills Training Session Quantity: 5; Behavioral: Family Skills Training Session Mode: Online; Behavioral: Family Skills Training Content: No Communication; Behavioral: Family Skills Training Content: No Cohesion
- Session 10, In-Person, Communication and Cohesion (Experimental): Participants will receive core behavioral weight loss group sessions and 10 family skills training sessions in-person with content covering communication and cohesion
  Interventions: Behavioral: Family Skills Training Session Mode: In-person; Behavioral: Family Skills Training Content: Communication; Behavioral: Family Skills Training Content: Cohesion; Behavioral: Family Skills Training Session Quantity: 10
- Session 10, In-Person, Communication and No Cohesion (Experimental): Participants will receive core behavioral weight loss group sessions and 10 family skills training sessions in-person with content covering communication but no cohesion
  Interventions: Behavioral: Family Skills Training Session Mode: In-person; Behavioral: Family Skills Training Content: Communication; Behavioral: Family Skills Training Session Quantity: 10; Behavioral: Family Skills Training Content: No Cohesion
- Session 10, In-Person, Cohesion and No Communication (Experimental): Participants will receive core behavioral weight loss group sessions and 10 family skills training sessions in-person with content covering cohesion but no no communication
  Interventions: Behavioral: Family Skills Training Session Mode: In-person; Behavioral: Family Skills Training Content: Cohesion; Behavioral: Family Skills Training Session Quantity: 10; Behavioral: Family Skills Training Content: No Communication
- Session 10, In-Person, No Communication and No Cohesion (Experimental): Participants will receive core behavioral weight loss group sessions and 10 family skills training sessions in-person with content covering no communication and no cohesion
  Interventions: Behavioral: Family Skills Training Session Mode: In-person; Behavioral: Family Skills Training Session Quantity: 10; Behavioral: Family Skills Training Content: No Communication; Behavioral: Family Skills Training Content: No Cohesion
- Session 10, On-Line, Communication and Cohesion (Experimental): Participants will receive core behavioral weight loss group sessions and 10 family skills training sessions on-line with content covering communication and cohesion
  Interventions: Behavioral: Family Skills Training Content: Communication; Behavioral: Family Skills Training Content: Cohesion; Behavioral: Family Skills Training Session Quantity: 10; Behavioral: Family Skills Training Session Mode: Online
- Session 10, On-Line, Communication and No Cohesion (Experimental): Participants will receive core behavioral weight loss group sessions and 10 family skills training sessions on-line with content covering communication but no cohesion
  Interventions: Behavioral: Family Skills Training Content: Communication; Behavioral: Family Skills Training Session Quantity: 10; Behavioral: Family Skills Training Session Mode: Online; Behavioral: Family Skills Training Content: No Cohesion
- Session 10, On-Line, Cohesion and No Communication (Experimental): Participants will receive core behavioral weight loss group sessions and 10 family skills training sessions on-line with content covering cohesion but no communication
  Interventions: Behavioral: Family Skills Training Content: Cohesion; Behavioral: Family Skills Training Session Quantity: 10; Behavioral: Family Skills Training Session Mode: Online; Behavioral: Family Skills Training Content: No Communication
- Session 10, On-Line, No Communication and No Cohesion (Experimental): Participants will receive core behavioral weight loss group sessions and 10 family skills training sessions on-line with content covering no communication and no cohesion
  Interventions: Behavioral: Family Skills Training Session Quantity: 10; Behavioral: Family Skills Training Session Mode: Online; Behavioral: Family Skills Training Content: No Communication; Behavioral: Family Skills Training Content: No Cohesion

INTERVENTIONS:
Behavioral: Family Skills Training Session Quantity: 5 — The number of family skills training sessions administered: 5 sessions
  Arms: Session 5, In-Person, Cohesion and No Communication; Session 5, In-Person, Communication and Cohesion; Session 5, In-Person, Communication and No Cohesion; Session 5, In-Person, No Communication and No Cohesion; Session 5, On-Line, Cohesion and No Communication; Session 5, On-Line, Communication and Cohesion; Session 5, On-Line, Communication and No Cohesion; Session 5, On-Line, No Communication and No Cohesion
Behavioral: Family Skills Training Session Mode: In-person — The mode of administration of family skills training sessions: in person or online
  Arms: Session 10, In-Person, Cohesion and No Communication; Session 10, In-Person, Communication and Cohesion; Session 10, In-Person, Communication and No Cohesion; Session 10, In-Person, No Communication and No Cohesion; Session 5, In-Person, Cohesion and No Communication; Session 5, In-Person, Communication and Cohesion; Session 5, In-Person, Communication and No Cohesion; Session 5, In-Person, No Communication and No Cohesion
Behavioral: Family Skills Training Content: Communication — The content of family skills training sessions administered focused on communication and conflict resolution : communication and conflict resolution
  Arms: Session 10, In-Person, Communication and Cohesion; Session 10, In-Person, Communication and No Cohesion; Session 10, On-Line, Communication and Cohesion; Session 10, On-Line, Communication and No Cohesion; Session 5, In-Person, Communication and Cohesion; Session 5, In-Person, Communication and No Cohesion; Session 5, In-Person, No Communication and No Cohesion; Session 5, On-Line, Communication and Cohesion; Session 5, On-Line, Communication and No Cohesion
Behavioral: Family Skills Training Content: Cohesion — The content of family skills training sessions administered focused on cohesion: cohesion or no cohesion
  Arms: Session 10, In-Person, Cohesion and No Communication; Session 10, In-Person, Communication and Cohesion; Session 10, On-Line, Cohesion and No Communication; Session 10, On-Line, Communication and Cohesion; Session 5, In-Person, Cohesion and No Communication; Session 5, In-Person, Communication and Cohesion; Session 5, In-Person, No Communication and No Cohesion; Session 5, On-Line, Cohesion and No Communication; Session 5, On-Line, Communication and Cohesion
Behavioral: Family Skills Training Session Quantity: 10 — The number of family skills training sessions administered: 10 sessions
  Arms: Session 10, In-Person, Cohesion and No Communication; Session 10, In-Person, Communication and Cohesion; Session 10, In-Person, Communication and No Cohesion; Session 10, In-Person, No Communication and No Cohesion; Session 10, On-Line, Cohesion and No Communication; Session 10, On-Line, Communication and Cohesion; Session 10, On-Line, Communication and No Cohesion; Session 10, On-Line, No Communication and No Cohesion
Behavioral: Family Skills Training Session Mode: Online — The mode of administration of family skills training sessions: online
  Arms: Session 10, On-Line, Cohesion and No Communication; Session 10, On-Line, Communication and Cohesion; Session 10, On-Line, Communication and No Cohesion; Session 10, On-Line, No Communication and No Cohesion; Session 5, On-Line, Cohesion and No Communication; Session 5, On-Line, Communication and Cohesion; Session 5, On-Line, Communication and No Cohesion; Session 5, On-Line, No Communication and No Cohesion
Behavioral: Family Skills Training Content: No Communication — The content of family skills training sessions administered focused on communication and conflict resolution : no communication and conflict resolution
  Arms: Session 10, In-Person, Cohesion and No Communication; Session 10, In-Person, No Communication and No Cohesion; Session 10, On-Line, Cohesion and No Communication; Session 10, On-Line, No Communication and No Cohesion; Session 5, In-Person, No Communication and No Cohesion; Session 5, On-Line, Cohesion and No Communication; Session 5, On-Line, No Communication and No Cohesion
Behavioral: Family Skills Training Content: No Cohesion — The content of family skills training sessions administered focused on cohesion: no cohesion
  Arms: Session 10, In-Person, Communication and No Cohesion; Session 10, In-Person, No Communication and No Cohesion; Session 10, On-Line, Communication and No Cohesion; Session 10, On-Line, No Communication and No Cohesion; Session 5, In-Person, Communication and No Cohesion; Session 5, On-Line, Communication and No Cohesion; Session 5, On-Line, No Communication and No Cohesion

SUMMARY:
The goal of this clinical trial is to learn the best combination of family components that yields optimal weight loss among Black adults. The main question it aims to answer is:

What combination of four family components in combination with a standard behavioral weight loss program yields optimal weight loss among Black adults? Researchers will compare different combinations of family skills components (communication content, cohesion content, number of sessions, and mode of delivery) to see the best weight loss.

Participants will:

* Participate in a 6-month behavioral weight loss intervention
* Attend core weight loss in-person group sessions, and dyad based family sessions
* Keep track of weight, dietary intake and physical activity

DETAILED DESCRIPTION:
This clinical trial aims to determine the most effective combination of family components to achieve optimal weight loss among Black adults. The main focus is to assess how different combinations of four family skills components-communication content, cohesion content, number of sessions, and mode of delivery-work together with a standard behavioral weight loss program.

Participants will engage in a 6-month behavioral weight loss intervention, which includes attending group weight loss sessions and family-based dyad sessions. They will also track their weight, dietary intake, and physical activity.

This is a 2 x4 factorial design with 16 study conditions.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as Black or African American (Index participant)
* BMI equal to greater than 30 kg/m^2 (Index); BMI equal to greater than 27.5 kg/m^2 (family partner)
* have a partner/family member willing to enroll in the study and must share a mutual goal of achieving weight loss
* English speaking
* ages 18-75
* any gender
* have access to and be able to use a smartphone, tablet, or computer that has web-access (this is required for data collection and some program components being tested)

Exclusion Criteria:

* participation in an intensive weight loss program (more than 12 visits) in the prior 6 months
* type 1 diabetes
* significant psychiatric illness, defined as depression or other major psychiatric illness not considered reasonably managed by counseling, medication, or both
* had bariatric surgery (surgery for weight loss) in the last 2 years or considering bariatric surgery in the next 6 months
* using or planning to start medications intentionally for weight loss
* are pregnant or planning to get pregnant in the next 6 months
* are breastfeeding and less than 2 months postpartum
* alcohol or substance abuse, defined as alcohol or substance use that interferes with work activities and/or has had a major negative impact on family/social function, the latter defined as more than 2 episodes per month.
* malignancy other than non-melanoma skin cancer, unless considered cured > 5 years ago. Exceptions include 1) men with localized prostate cancer (treated with usual modalities or managed with "active surveillance"), and 2) postmenopausal women receiving adjuvant endocrine therapy (e.g., aromatase inhibitor) for non-metastatic, hormone receptor-positive breast cancer
* self-report of advanced kidney disease (estimated glomerular filtration rate (GFR) < 30 mL/min)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body weight | baseline and 6 months
  Body weight (kg) expressed as a continuous variable will be collected on a digital scale.

SECONDARY OUTCOMES:
Mean Change in Blood Pressure | baseline and 6 months
  Both systolic and diastolic blood Pressure measured after 5 minutes of rest and taken in the same position throughout the study.
Change in skin carotenoids | baseline and 6 months
  To assess fruit and vegetable intake, skin carotenoids will be measured using a reflection spectroscopy device ("Veggie Meter") The Veggie Meter uses reflection spectroscopy and a light-emitting diode (LED) light to measure the skin's carotenoids on a scale of 0 to 800. Higher scores indicate more carotenoids, which usually means the person has eaten more fruits and vegetables.
Change in physical activity steps | baseline and 6 months
  To assess physical activity, the number of daily steps will be captured using a Fitbit wearable fitness tracker
Change in glycosylated hemoglobin (A1c) | baseline and 6 months
  Changes in A1c will be measured using a, Point of Contact A1c -Siemens Diabetes 5075 A1C Analyzer
Current Subjective Social Status | baseline
  Assesses a person's perceived rank relative to others in their group. The MacArthur Scale of Subjective Social Status (MacArthur SSS Scale) is a single-item measure that assesses a person's perceived rank relative to others in their group. Respondents view a drawing of a ladder with 10 rungs, and either read or hear that the ladder represents where people stand in society. Respondents further read or hear: "At the top of the ladder are the people who are the best off, those who have the most money, most education, and best jobs. At the bottom are the people who are the worst off, those who have the least money, least education, worst jobs, or no job. To score this measure, researchers simply note the number of the rung (1-10) on which the respondent placed their "X."
Change in Quality of Life | baseline and 6 months
  12-Item Short Form Survey (SF-12) assessing the impact of health on an individual's everyday life. The 12-Item Short Form Survey (SF-12) is scored by calculating two main scores: a Physical Component Summary (PCS) and a Mental Component Summary (MCS), both ranging from 0 to 100, with higher scores indicating better physical and mental health respectively
Change in Depression | baseline and 6 months
  Patient Health Questionnaire -8 (PHQ-8). To score the Patient Health Questionnaire-8 (PHQ-8), add up the scores from each of the eight items, with each item rated on a scale from 0 ("not at all") to 3 ("nearly every day") - resulting in a total score ranging from 0 to 24; higher scores indicate greater depression severity; generally, a score of 10 or higher is considered clinically significant for major depression, while scores between 5-9 are considered mild depression and 10-14 moderate depression.
Change in Perceived stress | baseline and 6 months
  Measured using Perceived Stress Scale 4 (PSS-4). On the Perceived Stress Scale 4 (PSS-4), each question is scored on a 0-4 scale, with higher scores indicating greater perceived stress, and the total score is calculated by adding up all four items; the possible score range for the PSS-4 is therefore 0-16, with higher scores signifying higher levels of stress.
Change for social support for exercise | baseline and 6 months
  The exercise participation subscale of the Social Support and Exercise Survey (10 items) measures social support specific to exercise behaviors. The subscale assesses the level of support for exercise from partners. Subscale example items include "Exercised with me" and "Criticized or made fun of me for exercising." Total scores range from 5 to 50, with higher scores indicating more social support for exercise participation behaviors.
Change in Self-Efficacy of Eating Behaviors | baseline and 6 months
  Measured by survey responses to the Weight Efficacy Lifestyle Questionnaire Short Form (WEL-SF).Scale goes from 0 (not at all confident) to 10 (very confident). Higher scores mean better self efficacy.
Change in Self-Efficacy of Physical Activity | baseline and 6 months
  The confidence subscale of the Patient-centered Assessment and Counseling for Exercise Adult Diet and Physical Activity Measure (6 items; ) measures confidence in participating in regular exercise or physical activity in different situations (e.g., "How confident are you that you would participate in regular exercise or physical activity: When I am tired?"). Items rated on a scale from 1 ("not at all confident") to 6 ("extremely confident"). Higher scores show higher self-efficacy.
Changes in self-regulation | baseline and 6 months
  Treatment Self-Regulation Questionnaire. To score the Treatment Self-Regulation Questionnaire (TSRQ), each item is typically rated on a 7-point Likert scale, where 1 represents "Not at all true" and 7 represents "Very true," with higher scores indicating a greater degree of autonomous motivation for engaging in the targeted health behavior;
Changes in nutrition self-efficacy | baseline and 6 months
  Nutrition Self-efficacy scale (5 items). To score a 5-item Nutrition Self-Efficacy scale, typically each item is rated on a Likert scale (usually 1-5, with 1 being "not at all confident" and 5 being "very confident"), and then the scores from all five items are added together to produce a total score, with higher scores indicating greater perceived self-efficacy in managing nutrition choices; the total score range would be between 5 (lowest self-efficacy) and 25 (highest self-efficacy)
Physical Activity Readiness | baseline
  PHYSICAL ACTIVITY READINESS QUESTIONNAIRE (PAR-Q) & You. The Physical Activity Readiness Questionnaire (PAR-Q) is a seven-question screening tool that helps determine if a person is healthy enough to exercise. If you answer "yes" to one or more questions, you should consult a physician before starting an exercise program
Change in Family Emotional Involvement | baseline and 6 months
  The family emotional involvement (7 items) of the Family Emotional Involvement and Criticism Scale rate items on a 5-point Likert scale, as above.
Change in Family Perceived Criticism | baseline and 6 months
  The perceived criticism (7 items) subscales of the Family Emotional Involvement and Criticism Scale rate items like on a 5-point Likert scale, as above.
Change in Family Collaborative problem solving | baseline and 6 months
  The Family Problem-Solving Communication Index (10 items) was used to measure the specific communication style that families use to manage and solve problems and conflicts in various types of stressful situations. Consisting of 2 subscales, affirmatory communication and incendiary communication, the response options were "false," "mostly false," "mostly true," and "true."
Change in Family Cohesion | baseline and 6 months
  The cohesion subscale (10 items) of the Family Adaptability and Cohesion Evaluation Scale III measures the emotional bonding family members have with one another. Items like "Family members ask each other for help" rated on a 5-point Likert scale from "almost never" to "almost always."
Personal Network Survey | baseline
  Social Network Analysis using Network Canvas software

OTHER OUTCOMES:
Change for social support for eating | baseline and 6 months
  The Social Support and Eating Habits Survey (10 items) measures social support specific to healthy eating. Subscales assess encouragement for eating behaviors from partners (e.g., "Encouraged me not to eat 'unhealthy food' when I am tempted") and discouragement for eating behaviors from partners (e.g., "Brought home foods I am trying not to eat"). The items are rated on a scale of "none" to "very often." Total scores range from 5 to 50, with higher scores indicating more social support for eating behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Samuel-Hodge, PhD, MS, RD, LDN, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to preserve all the study data and to make it available to other researchers as appropriate, except that audio recordings of semi-structured interviews will NOT be made available, but the transcripts of these interviews will be made available. We do not plan to transcribe the fidelity audio recordings, so these data will not be made available. Our rationale for not sharing the audio recorded data is to minimize the risk of loss of confidentiality. All stored data are de-identified. Data will be made available no later than the time of an associated publication.
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina.
Access Criteria: When data sharing is permitted, a Data Use Agreement (DUA) specifying the uses of such data to be shared must be in place before any data is shared. Requests can be submitted to the Industry Contracting for processing. The Principal Investigator must confirm that the DUA has been fully executed and IRB, IEC, or REB approval has been granted before sharing data.